CLINICAL TRIAL: NCT07384845
Title: The Role of Transcutaneous Vagus Nerve Stimulation in Neuroprotection and the Reduction of the Systemic Inflammatory Response in Acute Brain Injury
Brief Title: The Role of Transcutaneous Vagus Nerve Stimulation in Treatment of Acute Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Dinko Tonković, Professor Dinko Tonković, MD, PhD, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 02/013AG
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acute Brain Injury; Transcutaneous Vagus Nerve Stimulation; Neuromodulation; Immunomodulation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute brain injury patients with tVNS stimulation (Active Comparator): tVNS will be applied on left tragus, followed by stimulation with 20 Hz twice daily.
  Biomarkers of traumatic brain injury (S100B, neuron-specific enolase, GFAP), ghrelin and cytokine concentrations in serum and cerebrospinal fluid (IL-1β, IL-6, TNF-α, IL-10) will be measured on two occasions. CT angiography on the first and seventh day for patients with SAH.
  Interventions: Device: transcutaneous vagus nerve stimulation (tVNS)
- Acute brain injury patients with sham (Sham Comparator): tVNS VNS will be applied on left tragus, but without stimulation in the same time frame as in the first group. Biomarkers of traumatic brain injury (S100B, neuron-specific enolase, GFAP), ghrelin and cytokine concentrations in serum and cerebrospinal fluid (IL-1β, IL-6, TNF-α, IL-10) will be measured on two occasions. CT angiography on the first and seventh day for patients with SAH.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation (tVNS) — application of tVNS in patients with acute brain injury
  Arms: Acute brain injury patients with tVNS stimulation
Device: Sham (No Treatment) — TVNS will be placed in the same manner as in the first group, but without vagal stimulation
  Arms: Acute brain injury patients with sham

SUMMARY:
Acute brain injury is a major global health problem associated with high mortality and morbidity, limited therapeutic options, prolonged hospital stays, and long-term disability that significantly impairs quality of life and increases healthcare costs. Noninvasive transcutaneous VNS developed as a safer approach for treating cerebral edema, epileptic seizures, and blood-brain barrier disruption, for facilitating the recovery of motoric and cognitive functions, and for immunomodulation.

Transcutaneous VNS improves cerebral perfusion pressure and tissue oxygenation, supports reperfusion of the penumbral zone, and reduces neuronal hyperexcitability, thereby suppressing seizures.It may exert anti-inflammatory effects by reducing microglial cytokine and chemokine production. Additionally, vagal stimulation promotes acetylcholine-mediated suppression of pro-inflammatory cytokines, including TNF, IL-1β, IL-6, and IL-18.

Another anti-inflammatory mechanism involves ghrelin, a peptide hormone whose serum levels increase under vagal stimulation. Elevated ghrelin reduces TNF-α and other pro-inflammatory cytokines and may limit intracerebral hemorrhage by inhibiting the NLRP3 inflammasome and activating the Nrf2/ARE signaling pathway. Biomarkers such as S100 protein and neuron-specific enolase (NSE) are valuable indicators of brain tissue damage and clinical outcomes; tVNS may reduce their levels and support non-invasive monitoring of disease progression.

The technique is considered safe in patients .

To date, tVNS has not been evaluated in clinical trials in Croatia, nor reported in case studies or cohort analyses. Study outcomes will be correlated with patients' clinical status, duration and course of hospitalization, complication rates, and overall treatment outcomes.

DETAILED DESCRIPTION:
Acute brain injury is one of the leading health problems of today. It presents with high mortality and morbidity, limited therapeutic options, and prolonged hospital stays, leaving patients with disabilities that impair quality of life and increase healthcare costs. The etiology of brain injury may be traumatic or non-traumatic. The global incidence of traumatic brain injury (TBI) is estimated at 27 to 69 million cases per year, mainly due to falls and traffic accidents. Among the most challenging non-traumatic brain injuries is aneurysmal subarachnoid hemorrhage (aSAH), with an incidence of 10-15 patients per 100,000 per year. In the treatment of primary and secondary brain injury, both surgical and non-surgical procedures are important. Limited therapeutic options in the treatment of brain injury have opened the door to consideration of new non-invasive methods. Recent studies show that neuromodulation induced by vagus nerve stimulation (VNS) may contribute to better outcomes in patients with brain injury.

The first application of VNS in a clinical setting was an invasive procedure used in the treatment of pharmacoresistant epilepsy. Subsequently, a non-invasive method of transcutaneous VNS (tVNS) was developed, which may have neuroprotective and immunoprotective effects. According to existing research, tVNS provides a safer approach in the treatment of cerebral edema, epileptic seizures, disorders of the cerebral blood-brain barrier, recovery of motor and cognitive functions, and immunomodulation. Transcutaneous VNS induces enhanced regulation of endogenous noradrenergic activity through activation of the locus coeruleus and the release of noradrenaline in the amygdala, as well as higher overall concentrations of noradrenaline in the brain. Accordingly, an increase in cerebral perfusion pressure (CPP) enables better oxygenation of brain tissue and reperfusion of the penumbral zone. Noradrenaline suppresses seizures by protecting GABAergic neurons and reducing neuronal hyperexcitability. In addition, it exerts anti-inflammatory effects on microglial cells, reducing the production of cytokines and chemokines. Acetylcholine (ACh), under vagal stimulation, also reduces pro-inflammatory cytokines such as tumor necrosis factor (TNF), interleukins IL-1β, IL-6, and IL-18. At the same time, it influences the microglial phenotype, reducing the pro-inflammatory M1 microglial phenotype, which promotes oxidative stress and mitochondrial damage, in favor of the neuroprotective M2 phenotype. Recent studies show that tVNS also significantly modulates serum inflammatory cytokines in patients with sepsis. Another anti-inflammatory mechanism is the interaction of VNS with the peptide hormone ghrelin. Serum ghrelin concentrations increase under vagal stimulation, leading to a subsequent reduction in TNF-α levels and other pro-inflammatory cytokines after brain injury. Ghrelin also plays an important role in reducing intracerebral hemorrhage by inhibiting NLRP3 and stimulating the Nrf2/ARE signaling pathway. Analysis of biomarkers of brain tissue damage, such as S100 protein and neuron-specific enolase (NSE), can be used to assess mortality and morbidity, as well as outcomes of neurointensive care, and non-invasive tVNS stimulation could result in a reduction of their values and serve in monitoring the clinical condition of patients with brain injury.

Motor recovery depends on brain neuroplasticity, and the results of previous studies indicate significantly better functional motor recovery when rehabilitation therapy is combined with tVNS. Non-invasive tVNS can also alleviate cognitive dysfunction, as it reduces neuroinflammation and improves memory function through stimulation of peripheral and central cholecystokinin (CCK) receptors.

The use of tVNS is safe in patients with aSAH and stroke, and it significantly improves functional recovery in patients in a minimally conscious state after transauricular tVNS administered for a duration of four weeks.

To the best of our knowledge, tVNS has not yet been used in clinical trials in Croatia, nor has it been described in case reports or small cohort studies. The obtained results will be correlated with collected data on patients' clinical status, the course and duration of hospital treatment, the occurrence of complications, and treatment outcomes.

ELIGIBILITY:
IInclusion Criteria:

Patients over 18 years of age with a diagnosis of traumatic brain injury or acute subarachnoid hemorrhage due to rupture of an intracranial aneurysm, confirmed by brain CT or MRI.

Exclusion Criteria:

Patients under 18 years of age; patients with autoimmune diseases or malignant diseases; pregnant women; and patients for whom informed consent to participate in the study is not obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of traumatic brain injury (S100B, neuron-specific enolase, GFAP) and ghrelin | 7 days
  To measure and analyze the concentrations of biomarkers of traumatic brain injury (S100B, neuron-specific enolase [NSE], GFAP) as well as the peptide hormone ghrelin, in serum and cerebrospinal fluid within 24 hours of admission to the intensive care unit (ICU), and again after 7 days.
Cytokine concentrations in serum and cerebrospinal fluid (IL-1β, IL-6, TNF-α, IL-10) | 7 days
  To measure and analyze concentration of cytokines in serum and cerebrospinal fluid (IL-1β, IL-6, TNF-α, IL-10) within 24 hours of admission to the intensive care unit (ICU), and again after 7 days
CT angiography in patients with aneurysmatic SAH | 7 days
  Radiologically monitor the presence, development, and severity of vasospasm in patients with aSAH using CT angiography on two occasions: within 24 hours of the ruptured aneurysm closure, and on the 7th day after aneurysm closure

CONTACTS AND LOCATIONS:
Overall Officials: Dinko Tonković, Prof, MD PhD, Principal Investigator — Clinical Hospital Centre Zagreb; Martina Miklić Bublić, MD PhD, Principal Investigator — Clinical Hospital Centre Zagreb; Dunja Rogić, Prof, MD PhD, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- UHCZagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No